CLINICAL TRIAL: NCT00130091
Title: The Addition of Clonidine to 0.2% Ropivacaine for Wound Instillation After Minor Lower Abdominal Surgery in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital of Eastern Ontario (Other)
Responsible Party: Principal Investigator, Kimmo Murto, MD, FRCPC, Dept. Anesthesiology CHEO, Assistant Professor, University of Ottawa, Children's Hospital of Eastern Ontario
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 05/17E
Record Dates: First submitted 2005-08-11; First posted 2005-08-15 (Estimated); Last update posted 2015-02-20 (Estimated); Status verified 2015-02

CONDITIONS: Hernia, Inguinal; Hydrocele
Keywords: unilateral; hernia; hydrocele; pediatric; clonidine; nerve block
MeSH Terms: conditions — Hernia, Inguinal; Testicular Hydrocele; Hernia | interventions — Clonidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clonidine (Experimental): administer with local anesthetic
  Interventions: Drug: clonidine
- Local anesthetic (Placebo Comparator): Local anesthetic without clonidine
  Interventions: Drug: clonidine

INTERVENTIONS:
Drug: clonidine — 2 mcg clonidine added to local anesthetic

SUMMARY:
The current study will compare the effects on postoperative pain relief of "freezing" (ropivacaine 0.2 %) alone and in combination with clonidine for a nerve block in children undergoing hernia repair. The researchers anticipate that the addition of clonidine to "freezing" will result in prolongation of postoperative pain relief in children undergoing hernia repair compared to "freezing" used alone.

DETAILED DESCRIPTION:
The optimal method of controlling postoperative pain in children undergoing hernia repair would effectively relieve pain for extended periods of time and have no adverse effects. Unfortunately, such an ideal technique does not exist.

The control of postoperative pediatric pain after hernia repair is achieved with a combination of oral and intravenous pain medications and "nerve blocks". "Nerve blocks" are achieved by injecting local anesthetics or what is commonly referred to as "freezing "next to the nerve supply of the wound. "Freezing" the major nerves supplying sensation at the site of hernia repair in children, while they are asleep, is effective. At CHEO, this technique in addition to administering ketorolac, a liquid intravenous form of an anti-inflammatory agent similar to Advil, is the current technique of choice for postoperative pain control after inguinal hernia.

It is not unusual for these patients to require extra pain medications postoperatively. Available means of pain control in addition to those mentioned above include codeine-like medications, Tylenol, Advil-like medications and opioids administered intravenously. The addition of these medications increases the risk of suffering from side effects including respiratory depression, nausea and vomiting, and itching.

Ideally, the prolongation of postoperative pain relief by the addition of a second medication to the "freezing" during the nerve block would limit the need for additional pain medication and hence, decrease their associated side effects. Clonidine has the potential to be such a medication. It has been shown to provide pain relief by affecting several areas of the nervous system including the brain, the spinal cord and nerves. Clonidine prolongs pain relief of certain local anesthetics when used in nerve blocks for adults. Unfortunately, there are no studies that have examined the combination of clonidine and the local anesthetic ropivacaine for nerve blocks in children. Presently, the injectable form of clonidine is not marketed and is considered investigational in Canada.

The current study will be a prospective double -blind, randomized, controlled trial. It will compare the effects on postoperative pain relief of "freezing" (ropivacaine 0.2 %) alone and in combination with clonidine for a nerve block in children undergoing hernia repair. In addition, it will measure changes in the child's level of sedation, breathing, heart rate, blood pressure and any complications. Finally, it will assess how satisfied the parents are with this technique.

The researchers anticipate that the addition of clonidine to "freezing" will result in prolongation of postoperative pain relief in children undergoing hernia repair compared to "freezing" used alone.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral inguinal hernia or hydrocele
* 1 to 12 years old
* American Society of Anesthesiology classification I-II
* Written informed consent

Exclusion Criteria:

* Exclusion to nerve block
* Clotting disorder
* Infection
* Known allergy to clonidine or ropivacaine
* History of chronic, therapeutic administration of analgesics
* Receiving medications for attention deficit hyperactivity disorder
* Patients taking oral clonidine
* Undergoing bilateral hernia repair
* Morbid obesity

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2009-09; Primary Completion 2014-02 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Time to first analgesia after procedure | 24 hours

SECONDARY OUTCOMES:
continuous pain scores (modified Children's Hospital of Eastern Ontario Pain Score [mCHEOPS], modified Wong-Baker Faces) | baseline plus seven days
sedation scores | Between surgery and surgical day unit discharge (approx four hours)
emergence delirium score (Pediatric Anesthesia Emergence Delirium [PAED]) | Between surgery and surgical day unit discharge (approx four hours)
total analgesics consumed | seven days
total sedation consumed | Between surgery and surgical day unit discharge (approx four hours)

CONTACTS AND LOCATIONS:
Overall Officials: Kimmo Murto, MD, Principal Investigator — Children's Hospital of Eastern Ontario
Locations (1):
- Children's Hospital of Eastern Ontario, Ottawa, Ontario, Canada